CLINICAL TRIAL: NCT03166371
Title: Bioavailable Glutathione Supplementation: During Hospitalization and Beyond
Brief Title: Glutathione (GSH) Supplementation After Hospitalization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn prior to enrolling participants after being suspended due to funding and staffing issues.
Sponsor: Emory University (Other)
Collaborators: Your Energy Systems, LLC (Unknown)
Responsible Party: Principal Investigator, Thomas R. Ziegler, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00095819
Record Dates: First submitted 2017-05-12; First posted 2017-05-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Malnutrition
Keywords: Endocrinology; Nutrition; Aging
MeSH Terms: conditions — Malnutrition | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Glutathione (GSH) (Experimental): Participants will be randomized to receive two teaspoons containing 840 mg GSH (420 mg/tsp) twice daily for 90 days after discharge from Emory University Hospital (EUH).
  Interventions: Dietary Supplement: Liposomal Glutathione (GSH)
- Placebo (Placebo Comparator): Participants will be randomized to receive a placebo product identical to liposomal glutathione (GSH) twice daily for 90 days after discharge from Emory University Hospital (EUH).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Liposomal Glutathione (GSH) — Two teaspoons (containing 840 mg GSH, 420 mg/tsp) liposomal GSH (ReadiSorb®) will be taken orally twice daily for a total daily dose of 1680 mg GSH/day. Liposomal GSH will be refrigerated until use and mixed in ≈ 250 mL water or juice for oral intake. The study product will be consumed daily for 90 consecutive days after hospital discharge.
  Other Names: ReadiSorb®
  Arms: Liposomal Glutathione (GSH)
Other: Placebo — Two teaspoons of placebo product will be taken orally twice daily. The placebo will be refrigerated until use and mixed in ≈ 250 mL water or juice for oral intake. The placebo will be consumed daily for 90 consecutive days after hospital discharge.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if oral liquid glutathione treatment, has any effect on improving health-related cellular protection, muscle size and strength, and fatigue, weakness, and quality of life in older adults with a history of malnutrition who have been hospitalized. Persons enrolled in this study will be those initially admitted to Emory University Hospital (EUH) in Atlanta, GA, but recovering and ready to be discharged home or to an assisted living facility to eat an oral diet. A combination of nutritional measures, blood markers and imaging tools will assess body composition. Study participants will complete questionnaires about quality of life and physical health, and do simple testing for physical strength and stamina. Information from this pilot study will increase understanding of a simple intervention which may prevent or reduce health risks related to hospital recovery in older adults.

DETAILED DESCRIPTION:
This is a single-center randomized, double blind, placebo-controlled, intent-to-treat clinical trial to test the impact of oral administration of liposomal glutathione (GSH) in initially hospitalized, malnourished, older adults after discharge to the home setting. Study subjects will be clinically stable and able to complete serial study endpoint investigations. A total of 50 clinically stable subjects will be block-randomized to receive either oral liposomal GSH or identical placebo product for 90 days after discharge from Emory University Hospital (EUH). Plasma GSH redox status over time will be the primary study endpoint. Secondary study endpoints will include other thiol/disulfide indexes of oxidative stress, body composition, and measures of physical function, mobility, fatigue, frailty and quality of life. All endpoints will be determined at baseline (just prior to hospital discharge) and repeated at 30, 60 and 90 days after hospital discharge to the home or assisted living environment.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Emory University Hospital (EUH) and residing at home (including assisted living settings) before and after hospitalization
* Subject has voluntarily signed and dated an informed consent
* Greater than or equal to 5 and no more than 15 consecutive overnight stays in an Emory University Hospital general ward and/or Surgical Intensive Care Unit (SICU) or Medical Intensive Care Unit (MICU) during the current hospital admission
* Currently admitted to a general medical or surgical hospital ward at EUH and able to tolerate oral solid diet
* Positive screening prior to entry for mild, moderate or severe malnutrition by standard Centers for Medicare/Medicaid Services (CMS) criteria after hospital admission
* Currently mobile on hospital ward and able to be transported (wheelchair) to Clinical Research Unit for baseline testing
* Functionally ambulatory (self-reported ability to walk across a small room without assistance) during the 30 days prior to admission
* Ability to stand without assistance at the time of baseline testing
* Body mass index (BMI) >18.5, <40 mg/kg2
* Living within 40 miles of EUH

Exclusion Criteria:

* Subject not expected to be discharged to usual home or assisted living setting
* Requires tube feeding and/or parenteral nutrition in home/assisted living setting
* Planned or elective re-hospitalization within 90 days of discharge
* Inability to return to the EUH Clinical Research Unit for follow up study visits at 30, 60 and 90 days after entry into study
* History of acute or chronic gastrointestinal tract disorder that, in the opinion of the principal investigator would preclude ingestion or absorption of the study product (e.g., prior gastric bypass surgery, short bowel syndrome, inflammatory bowel disease, celiac disease, acute/chronic pancreatitis, or chronic upper gastrointestinal bleeding
* Current dementia, acute/chronic altered mental status, encephalopathy, brain metastases, eating disorders, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures in the opinion of the principal investigator
* History of stroke with motor disability or other significant movement disorders precluding protocol functional strength testing
* Acute hepatic failure during current hospitalization with total serum bilirubin > 3.5 mg/dL or transaminase values [alanine transaminase (ALT) and/or aspartate transaminase (AST) values > 3-fold the upper limit of normal range]
* Chronic or acute renal failure requiring chronic dialysis in home/assisted living setting after discharge
* Current active cancer or recently (within 6 months) treated cancer other than basal cell or squamous cell carcinoma of the skin or prostate cancer
* Participation in another research protocol within 30 days of entry into the current study or within 60 days after entry
* Any other condition or event considered exclusionary by the principal investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma Concentrations of GSH | Baseline, Post Hospital Discharge (90 Days)
  Plasma concentrations of GSH will be collected via blood draw.
Change in GSH/glutathione Disulfide (GSSG) Concentration Ratio | Baseline, Post Hospital Discharge (90 Days)
  GSH concentrations will be compared to glutathione disulfide. Concentrations will be collected and analyzed via blood draw.
Change in GSH/GSSH Pool Redox Potential (Eh) | Baseline, Post Hospital Discharge (90 Days)
  GSH and GSSH will be collected via blood draw. Redox potential is a measure of the tendency of a chemical species to acquire electrons and thereby be reduced. The more positive the potential, the greater the affinity for electrons and tendency to be reduced

SECONDARY OUTCOMES:
Body Composition assessed by Dual Energy X-ray Absorptiometry (DEXA) Scan | Baseline, Post Hospital Discharge (90 Days)
  The DEXA scan will assess body composition by defining lean body mass, total fat mass, and visceral fat mass.
Change in Waist Circumference | Baseline, Post Hospital Discharge (90 Days)
  Waist circumference will be measured in centimeters. Change is defined as the difference in measurements from baseline to 90 days post discharge.
Change in Hip Circumference | Baseline, Post Hospital Discharge (90 Days)
  Hip circumference will be measured in centimeters. Change is defined as the difference in measurements from baseline to 90 days post discharge.
Change in Body Mass Index (BMI) | Baseline, Post Hospital Discharge (90 Days)
  Body mass index (BMI) is a measure of body fat based on height and weight. A BMI below 18.5 = Underweight; 18.5 - 24.9 = Normal; 25.0 - 29.9 = Overweight; 30.0 and Above = Obese.
Change in Total Body Water (TBW) Volume | Baseline, Post Hospital Discharge (90 Days)
  Body water is the water content that is contained in the tissues, the blood, the bones and elsewhere. The average TBW% ranges for a healthy adult are: Females - 45 to 60%, Males - 50 to 65%.
Change in Intracellular Water Volume assessed by Bioelectrical Impedance Analysis (BIA) | Baseline, Post Hospital Discharge (90 Days)
  Intracellular water volume refers to water located within the cell. This will be measured by BIA, a method used for estimating body composition.
Change in Extracellular Water Volume assessed by Bioelectrical Impedance Analysis (BIA) | Baseline, Post Hospital Discharge (90 Days)
  Extracellular water volume refers to water located outside of the cell. This will be measured by BIA, a method used for estimating body composition.
Change in Phase Angle Measurements assessed by Bioelectrical Impedance Analysis (BIA) | Baseline, Post Hospital Discharge (90 Days)
  Phase angle is an indicator of cellular health and integrity. A low phase angle is consistent with an inability of cells to store energy and an indication of breakdown in the selective permeability of cellular membranes. A high phase angle is consistent with large quantities of intact cell membranes and body cell mass.
Change in Short Physical Performance Battery Score | Baseline, Post Hospital Discharge (90 Days)
  The Short Physical Performance Battery (SPPB) is a tool to assess lower extremity physical performance status.The scores range from 0 (worst performance) to 12 (best performance).
Change in Timed Up and Go Test Score | Baseline, Post Hospital Discharge (90 Days)
  The Timed Up and Go Test assesses mobility. Participants are asked to walk to a line 9.8 feet away, turn around at the line, and walk back at a normal pace. An older adult who takes ≥12 seconds to complete the TUG is at high risk for falling.
Change in Grip Strength assessed by Hand-Grip Dynamometry | Baseline, Post Hospital Discharge (90 Days)
  Handgrip Dynamometers are instruments for measuring the maximum isometric strength of the hand and forearm muscles, used for testing handgrip strength. Hand muscle measurements are as follows:
  Grade 5: full active range of motion & Normal muscle resistance Grade 4: full active range of motion & Reduced muscle resistance Grade 3: full active range of motion & No muscle resistance Grade 2: Reduced active range of motion & No muscle resistance Grade 1: No active range of motion & Palpable muscle contraction only Grade 0: No active range of motion & No palpable muscle contraction
Change in Life Space Assessment Questionnaire Score | Baseline, Post Hospital Discharge (90 Days)
  The Life Space Assessment Questionnaire assesses how much the person gets out and about and the spatial extent of the person's typical life space, i.e., what is the usual range of places in which the person engages in activities within the designated time frame.
Change in Iowa Fatigue Scale Score | Baseline, Post Hospital Discharge (90 Days)
  The Iowa Fatigue Scale assesses fatigue over the past month. General fatigue is a score between 30 and 39. Severe fatigue is a defined as a score between 40 - 55.
Change in Edmonton Frail Scale Score | Baseline, Post Hospital Discharge (90 Days)
  The Edmonton Frail Scale assesses and stratifies frailty. Scores range from 0-5 "not frail", 6-7 "vulnerable", 8-9 "mild frailty", 10-11 "moderate frailty", and 12-17 "severe frailty".
Change in Fatigue Symptom Inventory (FSI) Score | Baseline, Post Hospital Discharge (90 Days)
  The Fatigue Symptom Inventory (FSI), is a 14-item self-report measure designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life.
Plasma Concentrations of Cysteine (Cys) | Baseline, Post Hospital Discharge (90 Days)
  Plasma concentrations Cysteine (Cys) will be collected via blood draw.
Plasma Concentrations of Cistine (CySS) | Baseline, Post Hospital Discharge (90 Days)
  Plasma concentrations CySS will be collected via blood draw.
Cys/CySS Ratio | Baseline, Post Hospital Discharge (90 Days)
  Cys concentrations will be compared to CySS. Concentrations will be collected and analyzed via blood draw.
Cys/CySS Pool Redox Potential | Baseline, Post Hospital Discharge (90 Days)
  Cys and CySS will be collected via blood draw. Redox potential is a measure of the tendency of a chemical species to acquire electrons and thereby be reduced. The more positive the potential, the greater the affinity for electrons and tendency to be reduced

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University